CLINICAL TRIAL: NCT05692882
Title: To Evaluate the Safety and Efficacy of the NOVA Intracranial Drug-eluting Stent System in "real World" Patients with Intracranial Atherosclerotic Stenosis: a Prospective, Multicenter, Post-marketing Registry Clinical Study (NOVA II)
Brief Title: A Registry Study of Intracranial Atherosclerotic Stenosis Treatment by Intracranial Drug-eluting Stenting in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-NOVAII-202202
Record Dates: First submitted 2023-01-09; First posted 2023-01-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-03

CONDITIONS: Intracranial Arteriosclerosis; Stenosis Artery; Drug-Eluting Stents; Intracranial Artery Stenosis
Keywords: endovascular therapy; intracranial drug-eluting stent; symptomatic intracranial artery stenosis (sICAS)
MeSH Terms: conditions — Intracranial Arteriosclerosis | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Percutaneous transluminal angioplasty and stenting (Experimental): All patients will be implanted with Drug-Eluting Stents (NOVA DES).
  Interventions: Device: Drug-Eluting Stents

INTERVENTIONS:
Device: Drug-Eluting Stents — The NOVA stent is a sirolimus-eluting stent system designed for intracranial artery stenosis with a rapid exchangeable balloon

SUMMARY:
The primary objective of this trial is to evaluate the long-term safety and efficacy of the NOVA intracranial drug-eluting stent system in "real world" patients with intracranial atherosclerotic stenosis.

DETAILED DESCRIPTION:
The investigation is a prospective, multi-center, single arm clinical study. The trial is anticipated to last from December 2022 to December 2030 with 1000 subjects recruited in around 50 Chinese centers. The population for this study is subjects with intracranial atherosclerotic stenosis who are suitable candidates for stent angioplasty. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be enrolled after they signed the informed consent form. The study consists of ten visits including preoperative screening, operation date, 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years. The primary outcome was a composite of stroke or death within 30 days or any ischemic stroke or revascularization from the original culprit intracranial artery beyond 30 days through 12 months after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 80 years of age;
2. Symptomatic intracranial arteriosclerosis stenosis with reference diameter 2.25-4.00mm;
3. intracranial artery stenosis ( ≥70%) conformed by digital subtraction angiography (DSA);
4. Those who voluntarily participate in the study and sign informed consent form.

Exclusion Criteria:

1. Those who have surgery within previous 30 days or plan to perform major surgery in the next 90 days (surgery grade 3 and above);
2. Subjects of acute hemorrhagic stroke within 3 months;
3. The baseline mRS of disabling stroke is more than 3;
4. The target vessel is severely calcified and closely related to stenosis;
5. Non-atherosclerotic diseases (e.g. arterial dissection, Moya Moya disease, vascular inflammatory lesions caused by infection, autoimmune diseases, post-irradiation, postpartum status; developmental or genetic abnormalities such as fibromuscular dysplasia, sickle cell anemia, suspected vasospasm);
6. It is suspected that the ischemic event is due to embolism or arterial embolism from the extracranial segment (including ipsilateral chest or neck vascular occlusive disease) or potential cardiogenic embolism (e.g. atrial fibrillation, mitral stenosis, patent foramen ovale, left ventricular thrombus, myocardial infarction within 6 weeks, etc.);
7. Target artery's supplying artery stenosis > 50%. For example, patient with middle cerebral artery (MCA) severe stenosis (target artery) and the ipsilateral internal carotid artery (ICA) stenosis > 50% should be excluded; patient with basilar artery (BA) severe stenosis (target artery) and the dominant vertical artery (VA) stenosis > 50% should be excluded;
8. There are intracranial tumors, or intracranial arteriovenous malformations;
9. Those who are allergic to heparin, aspirin, clopidogrel, contrast agents, anesthetics, and stent components;
10. Pregnant and lactating women
11. Those who are unable to complete follow-up because of mental illness, cognitive or emotional disorders;
12. Inapplicable for this study at the investigators' viewpoints.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
stroke or death within 30 days or any ischemic stroke or revascularization from the original culprit intracranial artery beyond 30 days through 12 months after operation. | 1 year after operation
  The primary outcome was a composite of ischemic/hemorrhagic stroke and all-cause death within 30 days, or any ischemic stroke and revascularization from the original culprit intracranial artery beyond 30 days through 12 months after enrollment.

SECONDARY OUTCOMES:
Rate of any stroke (hemorrhagic/ischemic stroke) in the target blood supply area or all-cause death at 30 days after operation | 30 days after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke and any death in the target blood supply area
Rate of any stroke (hemorrhagic/ischemic stroke) in the non-target blood supply area or all-cause death at 30 days after operation | 30 days after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke and any death in the non-target blood supply area
Rate of transient ischemic attack at 30 days, 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  Transient ischemic attack (TIA) is a temporary blockage of blood flow to the brain with symptoms last from only a few minutes up to 24 hours
Rate of any stroke (hemorrhagic/ischemic stroke) in the target blood supply area at 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke in the target blood supply area
Rate of any stroke (hemorrhagic/ischemic stroke) in the non-target blood supply area at 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke in the non-target blood supply area
Rate of death (vascular/ non-vascular death) at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The cause of death was classified as vascular or nonvascular and based on information obtained from the family, medical records, and death certificates. Vascular death included death due to stroke, myocardial infarction (MI), heart failure, pulmonary embolus, cardiac arrhythmia, or other vascular cause.
Rate of symptomatic in-stent restenosis (ISR) and Revascularization at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  symptomatic ISR is defined as ISR associated with an ischemic event in the territory. Revascularization is the restoration or improvement of blood supply, and included surgical operation, endovascular procedures, etc.
Rate of modified Rankin Scale (mRS) at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
EuroQol-5D (EQ-5D) score at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  A health state defined by the descriptive EQ-5D system can be described by a five-digit number, each digit indicating the score of the corresponding dimension. For the description component a subject self-rates their health in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using either a three-level or a five-level scale.
Rate of in-stent restenosis at 1, 2, 3, 4 years and 5 years after operation (Optional) | 1, 2, 3, 4 years and 5 years after operation
  Patients with ≥50% stenosis of the vessel
Rate of Device defect | within 5 years of whole trial
  Device defects refer to the unreasonable risks that may endanger human health and life safety during the normal use of medical devices in the course of clinical trials, such as label errors, quality problems, failures, etc.
Rate of bleeding events at 1 years after operation | 1 year after operation
  Bleeding was defined according to Bleeding Academic Research Consortium

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Zhongrong, Principal Investigator — Beijing Tiantan Hospital
Locations (5):
- China (5):
  - First People's Hospital of Chenzhou, Chenzhou
  - Ganzhou People's Hospital, Ganzhou
  - Jinhua Municipal Central Hospital, Jinhua
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Shanxi Cardiovascular Hospital, Shanxi